CLINICAL TRIAL: NCT06943638
Title: The Effect of Mild Exercise While Receiving Chemotherapy on the Psychology of the Cancer Patient
Brief Title: How Easy-to-Follow Exercises Can Help Cancer Patients With Anxiety While Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christine Mavrogiannopoulou (Other)
Responsible Party: Sponsor-Investigator, Christine Mavrogiannopoulou, Clinical Researcher, University of Crete
Organization: University of Crete (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 779/15-1-2024
Record Dates: First submitted 2025-03-24; First posted 2025-04-24 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Exercise; Stress
Keywords: cancer; physiotherapy; exercise; physical therapy; chemotherapy; stress
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild exercise and stretching (Experimental): They received individualized workout and stretching programme to relieve some of the stress
  Interventions: Other: Mild Exercise and stretches

INTERVENTIONS:
Other: Mild Exercise and stretches — For 15 minutes the patient received an individualized mild workout program intending to relax and relieve some of his stress. The workout includes deep breaths, easy-to-do exercises, and stretches from lying on the bed, sitting in a chair, or standing. I always followed the patient's tempo and provided him with as many breaks as he needed.

SUMMARY:
Cancer is one of the main causes of death, and this study looks at how light exercise and stretching might reduce anxiety in patients receiving chemotherapy. The research took place in a hospital's daily care unit and used a study design where each patient was compared to themselves, measuring anxiety before and after the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) with cancer receiving chemotherapy
* Signed patient consent

Exclusion Criteria:

* The denial of the patient
* The occurrence of side effects from the treatment (such as dizziness, nausea, severe fatigue)
* Patients with low cognitive level where they could not follow simple instructions
* Patients with hearing disorders that prevented them from following simple instructions
* Patients who could not mobilize independently.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- General Oncological Hospital of Kifisia Oi Agioi Anargyroi, Athens, Kifissia, Greece

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because this research doesn't require the reproduction of special types of patients. They need to have cancer, receive chemotherapy, and be adults.

REFERENCES:
- [Background] Furmaniak AC, Menig M, Markes MH. Exercise for women receiving adjuvant therapy for breast cancer. Cochrane Database Syst Rev. 2016 Sep 21;9(9):CD005001. doi: 10.1002/14651858.CD005001.pub3. PMID 27650122
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the General Oncology Hospital of Kifissia "Agioi Anargyroi" in Athens, Greece. Eligible patients undergoing chemotherapy were invited to participate during routine clinical visits. Written informed consent was obtained from all participants.
Pre-assignment Details: There are no pre-assignement details
Period: Overall Study
Arm/Group | Mild Exercise and Stretching
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants (N=45) were included in the baseline analysis.
Arm/Group | Mild Exercise and Stretching
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] — The age was calculated by the year of birth
  Years | 68.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants] — We only accepted male or female as sex of the participants
  Participants
    Female | 20
    Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants] — All participnts were enrolled from the Greek oncological Hospital in Kifissia, Athens
  Participants
    Greece | 45

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Anxiety Assessment Scale (STAI-State) for Cancer Patients Receiving Chemotherapy Doing Mild Exercises and Stretches
Description: The STAI-State (Greek version, State-Trait Anxiety Inventory -STAI-) will be used to assess anxiety levels in cancer patients undergoing chemotherapy, before and after a brief exercise intervention. The STAI-State scale has a 20-item questionnaire where individuals rate how they feel at a particular moment on a scale from "not at all" to "very much so." "Not at all" equal to 1, "Somewhat" to 2, "Moderately so" to 3, "Very much so" to 4. Scores are submitted and range from 20 to 80, with higher scores indicating greater anxiety. No subscale is required to compute At baseline (Time = 0 minutes), participants complete the STAI-State scale. They then engage in a 15-minute mild exercise and stretching program tailored to their physical condition. In some cases, particularly among younger participants, the session may be conducted in small groups of up to 2 individuals. Immediately post-intervention (approximately 20 minutes from baseline), participants complete the STAI-State scale again.
Time Frame: Baseline and approximately 20 minutes post-intervention
Measure: Mean (Standard Deviation); unit: STAI-State score
Arm/Group | Mild Exercise and Stretching
Number analyzed (Participants) | 45
STAI-State score
  Pre- intervention | 37.73 (13.33)
  Post- intervention | 32 (14.22)
Statistical Analysis 1: Comparison: Mild Exercise and Stretching; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: from enrollment until the end of exercise, up to 20 minutes
Description: no adverse events reported
Arm/Group | Mild Exercise and Stretching
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
The small sample size (n=45) limits generalizability. All participants came from one hospital's Day Care Unit in northern Athens, introducing selection bias. The single 20-minute session and no follow-up restrict conclusions on long-term effects. Including various cancer types without stratified analysis adds heterogeneity. No control group and reliance on self-reports may bias results. Many declined participation due to fatigue or unfamiliarity with exercise.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT06943638/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT06943638/SAP_001.pdf
  • Informed Consent Form: document to inform patients about the process (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT06943638/ICF_002.pdf